CLINICAL TRIAL: NCT04860882
Title: HEart Surgery In Atrial Fibrillation and Supraventicular Tachycardia
Acronym: HEIST
Status: Completed | Type: Observational
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Mariusz Kowalewski, PhD, M.D., Nicolaus Copernicus University
Other Study IDs: HEIST
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, heart surgery, cabg, valve surgery, preoperative, mortality, grafts
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation is the most common cardiac arrhythmia, the incidence of which increases drastically with age. As more and more elderly patients undergo heart surgery, the proportion of patients in this population will increase. Atrial fibrillation has been shown to be a poor prognostic factor in several surgical situations. The aim of our study was to assess long-term mortality among patients with preoperative AF under various cardiac surgery settings, with a particular emphasis on the strategy of coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Referred for heart surgery,
* preoperative atrial fibrillation

Exclusion Criteria:

* age<18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation referred for cardiac surgery in the 5 Polish participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Death from any cause | 2008-2020
  Through polish national health fund we are able to determine patient status (dead or alive)